CLINICAL TRIAL: NCT02764892
Title: An Open Label Study of V81444 Using Positron Emission Tomography to Assess Occupancy of Brain Adenosine A2A Receptors & Functional & Perfusion MRI to Explore Effects on Regional Brain Activity & Perfusion in Healthy Male Volunteers
Brief Title: A Study in Healthy Male Volunteers to Investigate a New Drug for the Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vernalis (R&D) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: V81444-1PD-02
Record Dates: First submitted 2015-09-25; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- V81444 (Experimental): Single oral dose of V81444
  Interventions: Drug: V81444

INTERVENTIONS:
Drug: V81444 — Single oral dose of V81444

SUMMARY:
The main purpose of the study is to identify the best dose of V81444 to use in future trials in patients with Parkinson's disease. The study will also explore the effects of V81444 on brain activity and blood flow with tests of mental ability ("cognitive function tests"). It will also check how safe V81444 is and how well it is tolerated after dosing.

DETAILED DESCRIPTION:
In this Phase I, single-centre, open-label, adaptive, single-dose study at multiple dose levels, the relationship between dose and plasma concentration of orally administered V81444 to brain A2A RO was investigated in 6 healthy male volunteers. In addition, the effects of V81444 on regional brain activity and perfusion during tests of cognitive function, and the safety and tolerability of V81444 were assessed. For each subject, the study consisted of a screening visit, a baseline visit, a treatment period, and a safety follow-up visit. The dose of V81444 and timing of scans performed were defined in the protocol for the first 2 subjects only. The dose, nature and timings of assessments for subsequent subjects were determined based on review of emerging receptor binding, pharmacokinetic (PK), pharmacodynamic (PD) and safety information.

In each treatment period, subjects were admitted to the unit on the day before dosing (Day -1), received a single oral dose of V81444 on Day 1 and, subject to satisfactory medical review, were discharged a minimum of 12 h after dosing. Overall, 3 doses of V81444 were assessed (250 mg, 50 mg, and 100 mg), with 2 subjects included at each dose level. PD assessments were performed at baseline and after each dose of V81444 using PET (with the A2A radioligand, to measure brain A2A RO, as well as MRI techniques to investigate the effects of V81444 on regional brain activity and perfusion during cognitive function tests. PK parameters were assessed by assay of V81444 concentration in plasma. Safety and tolerability were assessed by monitoring physical examination findings, adverse events (AEs), vital signs, 12 lead electrocardiogram (ECG) and clinical laboratory safety tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers: aged 25 to 55 years, in good general health as determined by medical history, physical examination and screening investigations, and taking no regular medication.
* Confirmation to be sought for all volunteers that their general practitioner has provided an acceptable medical history.

Exclusion Criteria:

* Any significant medical condition or a history of such a condition that the Investigator considers should exclude the subject from the study.

Specific exclusion criteria relate to

* usual caffeine intake and willingness to abstain from caffeine
* history or evidence of clinically significant gastro-intestinal disease
* presence of structural brain abnormality
* contraindications or cautions for MRI scanning
* clotting test results
* exposure to significant levels of ionising radiation in the past

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentration V81444 corresponding with 50% brain A2A receptor occupancy. | Up to 27 hours after a single dose
  Plasma concentrations of V81444 and binding of [11C]SCH442416 radioligand to brain A2A receptors using PET before and after V81444 dosing to determine occupancy of A2A receptors by V81444.

SECONDARY OUTCOMES:
Cognitive function using functional MRI | 5 hours after dosing
Change versus placebo in proportion of subjects with adverse events | Up to 7 Days after last dose
Change versus placebo in proportion of subjects with abnormal laboratory findings | Up to 7 Days after last dose
Change versus placebo in proportion of subjects with clinically significant abnormalities on vital signs | Up to 7 Days after last dose
Change versus placebo in proportion of subjects with clinically significant abnormalities in 12-lead ECG | Up to 7 Days after last dose
Change versus placebo in proportion of subjects with clinically significant abnormalities on physical examination | Up to 7 Days after last dose